CLINICAL TRIAL: NCT01738568
Title: Effect of Aging and Aerobic Exercise Training on Brain Glucose Metabolism
Brief Title: Effects of Aging and Aerobic Exercise Training on Brain Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Val Lowe, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-003357
Record Dates: First submitted 2012-11-27; First posted 2012-11-30 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Dementia
Keywords: High intensity aerobic training
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Aerobic exercise
  Interventions: Behavioral: High intensity aerobic training; Behavioral: Sedentary Control

INTERVENTIONS:
Behavioral: High intensity aerobic training — High intensity aerobic interval training will be performed 12-weeks. Exercise training will last 1 hour per day, 5 days per week and include high intensity interval cycling at ~70-95% maximum workload for 4 minutes followed by 3 minutes of rest.
Behavioral: Sedentary Control — Sedentary control participants will not perform any regular exercise for 12-weeks.

SUMMARY:
Aging is associated with a loss of brain function and conditions such as dementia and Alzheimer's disease. It is likely that decreased brain metabolism is contributing to the progression of age related degenerative diseases. Aerobic exercise training can increase brain volumes and is associated with decreased risk for degenerative brain conditions. However, little is know about the changes that occur to brain metabolism with aerobic training and aging.

ELIGIBILITY:
Healthy sedentary adults aged 18-30 or 65-80 years of all ethnicities will be eligible. Pregnant women, children, prisoners or other at risk populations will not be recruited.

Inclusion Criteria:

* Age 18-30 years or 65-80 years

Exclusion Criteria:

* Body mass index (BMI) >31 kg/m2
* Smoking
* Pregnancy
* Participation in structured exercise (>2 times per week for 30 minutes or longer)
* Cardiovascular, metabolic (type 2 diabetes, fasting plasma glucose at or above 110 mg/dL and untreated hypo- or hyperthyroidism) or renal disease
* Orthopedic problems that would keep them from being able to ride an exercise bicycle, lift weights or do a combination of these exercise
* Medications that are known to impact on mitochondrial function: Corticosteroids, opiates, benzodiazepines, tricyclic antidepressants, beta blockers, sulfonylureas, insulin, anticoagulants, barbiturates, insulin sensitizers, fibrates (PPAR gamma agonist)
* Claustrophobia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-10; Primary Completion 2015-02-12 (Actual); Study Completion 2015-02-12 (Actual)

PRIMARY OUTCOMES:
Change in Brain Glucose Uptake | 12 weeks
  The investigators will assess brain glucose uptake using positron emission tomography at baseline and following 12-weeks of either aerobic exercise training or sedentary control period.

CONTACTS AND LOCATIONS:
Overall Officials: Val Lowe, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Robinson MM, Lowe VJ, Nair KS. Increased Brain Glucose Uptake After 12 Weeks of Aerobic High-Intensity Interval Training in Young and Older Adults. J Clin Endocrinol Metab. 2018 Jan 1;103(1):221-227. doi: 10.1210/jc.2017-01571. PMID 29077855
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials